CLINICAL TRIAL: NCT01814176
Title: Measurement of Forces Applied Using a Macintosh Direct Laryngoscope Compared to GlideScope Video Laryngoscope in Patients With at Least One Difficult Intubation Risk Factor
Brief Title: Measurement of Forces Applied Using a Macintosh Direct Laryngoscope Compared to GlideScope Video Laryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-0229-B
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2013-03

CONDITIONS: Moderately Difficult to Intubate
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Macintosh Direct Laryngoscope (Active Comparator): 2 main forces - a 'lifting' force to elevate the structures not in the line of sight and a force exerted by the user's wrist to counterbalance the torque effect of the tongue tissues on the blade
  Interventions: Device: Intubation with GlideScope Video Laryngoscope or Macintosh Direct Laryngoscope
- GlideScope Video Laryngoscope (Active Comparator): The GlideScope has a 60º angulation anteriorly at the distal portion of the blade, allowing an anterior view of the larynx.
  Interventions: Device: Intubation with GlideScope Video Laryngoscope or Macintosh Direct Laryngoscope

INTERVENTIONS:
Device: Intubation with GlideScope Video Laryngoscope or Macintosh Direct Laryngoscope

SUMMARY:
During Anesthesia many patients require that a breathing be inserted into their windpipe. This is usually achieved using a direct laryngoscope, consisting of a retraction blade with a light near its end. When achieving a direct line-of-sight to the windpipe is difficult, more force is often applied, resulting in greater patient stress. A GlideScope video laryngoscope uses a camera and light source to see the windpipe. This enables the user to see objects that may not be in the direct line-of-sight. This likely results in less force being required, reducing patient stress. Because such stresses are often confounded by patient variables, we are comparing the forces required by the direct and video laryngoscopes on patients with at least one risk factor for difficulty, by directly measuring these with special sensors attached to the laryngoscope blades.

ELIGIBILITY:
Inclusion Criteria:

* age > 18years
* elective surgery
* single lumen endotracheal intubation required
* signed informed consent
* one risk factor for a difficult laryngoscopy ( Mallampati score >3, inter-incisor gap < 3.5cm, thyromental distance < 6.5cm, sternomental distance < 12.5cm, reduced neck extension and flexion)

Exclusion Criteria:

* lack of patient consent
* anesthesiologist declines to consent
* contraindication to neuromuscular blockade
* ASA 4
* rapid sequence intubation
* previous failed intubation
* other method of intubation indicated eg fiberoptic intubation, awake tracheostomy
* symptomatic gastro-esophageal reflux
* cervical spine instability
* unstable hypertension and symptomatic coronary artery disease
* cerebrovascular disease or raised intracranial pressure
* oral/pharyngeal/laryngeal carcinoma
* loose teeth/poor dentition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Peak forces during intubation | Intraoperatively
  Peak forces generated during the laryngoscopy and intubation process using both laryngoscopes.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Cordovani D, Russell T, Wee W, Suen A, Cooper RM. Measurement of forces applied using a Macintosh direct laryngoscope compared with a Glidescope video laryngoscope in patients with predictors of difficult laryngoscopy: A randomised controlled trial. Eur J Anaesthesiol. 2019 Mar;36(3):221-226. doi: 10.1097/EJA.0000000000000901. PMID 30308524